CLINICAL TRIAL: NCT03801135
Title: A Prospective Interventional Study to Investigate Changes in Haemostasis After Therapeutic Plasmapheresis With Citrate Anticoagulation With or Without Coagulation Factors Replacement
Brief Title: Changes in Haemostasis After Therapeutic Plasmapheresis With Citrate Anticoagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matej Zrimsek, Principal Investigator, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MPFhemostaza
Record Dates: First submitted 2018-10-04; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Humoral Rejection; Guillain-Barre Syndrome; Miller Fisher Syndrome; CIDP; Good Pasture Syndrome; Hyperviscosity Syndrome
Keywords: Fibrinogen concentrate; Fresh frozen plasma; ROTEM; Fibrinogen; Overall coagulation potential
MeSH Terms: conditions — Guillain-Barre Syndrome; Miller Fisher Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Anti-Glomerular Basement Membrane Disease | interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrolyte&Albumin Group (No Intervention): One calculated plasma volume will be replaced with a mixture of electrolyte replacement solution and albumin.
- Fibrinogen Treatment Group (Experimental): One calculated plasma volume will be replaced with a mixture of electrolyte replacement solution and albumin. Fibrinogen concentrate will be infused afterwards.
  Interventions: Drug: Fibrinogen concentrate
- FFP Treatment Group (Active Comparator): One calculated plasma volume will be replaced with a mixture of electrolyte replacement solution, albumin and fresh frozen plasma.
  Interventions: Other: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Fibrinogen concentrate — Haemocomplettan will be infused after plasma exchange procedure
  Other Names: Haemocomplettan
  Arms: Fibrinogen Treatment Group
Other: Fresh Frozen Plasma — Fresh frozen plasma will be part of replacement fluid
  Arms: FFP Treatment Group

SUMMARY:
Plasma exchange procedures remove procoagulant and anticoagulant factors. Every procedure increases the risk of bleeding and repeated procedures increase the risk of bleeding mostly because lower fibrinogen levels. The aim of study is to define coagulation status of patient after plasmapheresis with different laboratory tests and to investigate the possibility of fibrinogen concentrate replacement for the correction of induced coagulation disorder.

ELIGIBILITY:
Inclusion Criteria:

* Every patient who will need repeated plasmapheresis treatment in UKC Ljubljana

Exclusion Criteria:

* pregnancy
* coagulation disorders
* Hypertriglyceridemia-induced acute pancreatitis
* hepatic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-24 (Estimated)

PRIMARY OUTCOMES:
Effect of plasmapheresis replacement fluid type on fibrinogen level | Right after every plasmapheresis session, during the whole plasmapheresis treatment (usually about 2 weeks)]
  Change of fibrinogen level after plasmapheresis treatment depending on replacement fluid type

SECONDARY OUTCOMES:
Effect on coagulation tests after plasmapheresis - ROTEM EXTEM | Right after every plasmapheresis session, during the whole plasmapheresis treatment (usually about 2 weeks)]
  ROTEM (EXTEM MCF) change after plasmapheresis treatment depending on replacement fluid type
Effect on coagulation tests after plasmapheresis - ROTEM FIBTEM | Right after every plasmapheresis session, during the whole plasmapheresis treatment (usually about 2 weeks)]
  ROTEM (FIBTEM MCF) change after plasmapheresis treatment depending on replacement fluid type

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Gorenjska, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zrimsek M, Gubensek J, Marn Pernat A. A Pilot Study on the Replacement of Fibrinogen with Fibrinogen Concentrates During Therapeutic Plasma Exchange with Mild to Moderate Bleeding Risk-A Comparison with Fresh Frozen Plasma and Albumin Replacement. J Clin Med. 2024 Dec 16;13(24):7662. doi: 10.3390/jcm13247662. PMID 39768590